CLINICAL TRIAL: NCT04481750
Title: Phase I Study of Oral Edaravone in Healthy Adult Males (Single- and Multiple-dose Study)
Brief Title: Study of Oral Edaravone in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MT-1186-J01
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- A single dose MT-1186 (Part 1, Cohort S1) (Experimental): Healthy Japanese male subjects receive a single dose of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- A single dose MT-1186 (Part 1, Cohort S2) (Experimental): Healthy Japanese male subjects receive a single dose of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- A single dose MT-1186 (Part 1, Cohort S3-1) (Experimental): Healthy Japanese male subjects receive doses of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- A single dose MT-1186 (Part 1, Cohort S3-2) (Experimental): Healthy Japanese male subjects receive doses of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- A single dose MT-1186 (Part 1, Cohort S4) (Experimental): Healthy Japanese male subjects receive a single dose of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- A single dose MT-1186 (Part 1, Cohort S5) (Experimental): Healthy Japanese male subjects receive a single dose of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- A single dose MT-1186 (Part 1, Cohort S6) (Experimental): Healthy Japanese male subjects receive a single dose of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- A single dose MT-1186 (Part 1, Cohort S7) (Experimental): Healthy Caucasian male subjects receive a single dose of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- Multiple doses MT-1186 (Part 2, Cohort M1) (Experimental): Healthy Japanese male subjects receive multiple doses of MT-1186 or matching placebo.
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo
- Multiple doses MT-1186 (Part 2, Cohort M2) (Experimental): Healthy Japanese male subjects receive multiple doses of MT-1186 or matching placebo
  Interventions: Drug: MT-1186; Drug: MT-1186-matching placebo

INTERVENTIONS:
Drug: MT-1186 — Solution or suspension
  Other Names: Edaravone
Drug: MT-1186-matching placebo — Solution or suspension

SUMMARY:
To evaluate the pharmacokinetics safety, and tolerability of single and multiple doses of edaravone solution and suspension in healthy adult males

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* Healthy adult male volunteers
* Japanese or Caucasian
* Subjects aged between 20 and 45 years at the time of informed consent
* Subjects who have thoroughly understood the contents of the study and voluntarily provided written informed consent to participate in the study

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Subjects with a current or previous history of cardiac, hepatic, renal, gastrointestinal, respiratory, psychiatric/nervous, hematopoietic, or endocrine diseases, and those whom the investigator (or subinvestigator) deems unsuitable for the study
* Body mass index (BMI) of <18.0 or >30.0, or body weight of <50 kg (BMI formula: body weight [kg]/height [m]2, rounded to one decimal place)
* Subjects who have undergone any surgery known to affect the gastrointestinal absorption of drugs
* Subjects who do not agree to use an effective method of contraception from initiation of study drug administration to 14 days after completion (discontinuation) of study drug administration
* Subjects who have previously received edaravone
* Subjects who have participated in another clinical study and received a study drug within 12 weeks before providing informed consent

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (1):
- Investigational Site, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shimizu H, Nishimura Y, Shiide Y, Matsuda H, Akimoto M, Matsuda M, Nakamaru Y, Kato Y, Kondo K. Evaluation of Pharmacokinetics, Safety, and Drug-Drug Interactions of an Oral Suspension of Edaravone in Healthy Adults. Clin Pharmacol Drug Dev. 2021 Oct;10(10):1174-1187. doi: 10.1002/cpdd.925. Epub 2021 Mar 11. PMID 33704925
- [Derived] Shimizu H, Nishimura Y, Shiide Y, Akimoto M, Matsuda H, Kato Y, Hirai M. Food Effect Study to Assess the Impact on Edaravone Pharmacokinetic Profiles in Healthy Participants. Clin Ther. 2022 Dec;44(12):1552-1565. doi: 10.1016/j.clinthera.2022.10.001. Epub 2022 Nov 12. PMID 36376130

RESULTS

PARTICIPANT FLOW:
Groups:
- A Single Dose MT-1186 (Part 1, Cohort S1): Healthy Japanese male subjects receive a single dose of MT-1186 60 mg solution.
- A Single Dose MT-1186 (Part 1, Cohort S2): Healthy Japanese male subjects receive a single dose of MT-1186 120 mg suspension.
- A Single Dose MT-1186 (Part 1, Cohort S3): Healthy Japanese male subjects receive a single dose of MT-1186 200 mg under fasted condition in period 1, and fed condition in period 2 with washout period at least 4-day.
- A Single Dose MT-1186 (Part 1, Cohort S4): Healthy Japanese male subjects receive a single dose of MT-1186 300 mg suspension with xanthan.
- A Single Dose MT-1186 (Part 1, Cohort S5): Healthy Japanese male subjects receive a single dose of MT-1186 300 mg suspension.
- A Single Dose MT-1186 (Part 1, Cohort S6): Healthy Japanese male subjects receive a single dose of MT-1186 30 mg suspension.
- A Single Dose MT-1186 (Part 1, Cohort S7): Healthy Caucasian male subjects receive a single dose of MT-1186 200 mg suspension.
- Matching Placebo (a Single Dose Cohorts): Healthy Japanese/Caucasian male subjects receive a single dose of matching placebo.
- Multiple Doses MT-1186 (Part 2, Cohort M1): Healthy Japanese male subjects receive multiple doses of MT-1186 120 mg suspension.
- Multiple Doses MT-1186 (Part 2, Cohort M2): Healthy Japanese male subjects receive multiple doses of MT-1186 200 mg suspension.
- Matching Placebo (Multiple Doses Cohorts): Healthy Japanese male subjects receive multiple doses of matching placebo.
Period: Period 1 (Fasted)
Arm/Group | A Single Dose MT-1186 (Part 1, Cohort S1) | A Single Dose MT-1186 (Part 1, Cohort S2) | A Single Dose MT-1186 (Part 1, Cohort S3) | A Single Dose MT-1186 (Part 1, Cohort S4) | A Single Dose MT-1186 (Part 1, Cohort S5) | A Single Dose MT-1186 (Part 1, Cohort S6) | A Single Dose MT-1186 (Part 1, Cohort S7) | Matching Placebo (a Single Dose Cohorts) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2) | Matching Placebo (Multiple Doses Cohorts)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 6 | 6 | 6
Completed | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 14 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (After Meal)
Arm/Group | A Single Dose MT-1186 (Part 1, Cohort S1) | A Single Dose MT-1186 (Part 1, Cohort S2) | A Single Dose MT-1186 (Part 1, Cohort S3) | A Single Dose MT-1186 (Part 1, Cohort S4) | A Single Dose MT-1186 (Part 1, Cohort S5) | A Single Dose MT-1186 (Part 1, Cohort S6) | A Single Dose MT-1186 (Part 1, Cohort S7) | Matching Placebo (a Single Dose Cohorts) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2) | Matching Placebo (Multiple Doses Cohorts)
Started | 0 (This cohort was closed in Period 1) | 0 (This cohort was closed in Period 1) | 5 (Cohort S3 is a crossover study consisting of Period 1 (Cohort S3-1) and Period 2 (Cohort S3-2). Out of 6 subjects, only 5 subjects received MT-1186 in COhort S3-2.) | 0 (This cohort was closed in Period 1) | 0 (This cohort was closed in Period 1) | 0 (This cohort was closed in Period 1) | 0 (This cohort was closed in Period 1) | 0 (This cohort was closed in Period 1) | 0 (This cohort was closed in Period 1) | 0 (This cohort was closed in Period 1) | 0 (This cohort was closed in Period 1)
Completed | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Single Dose MT-1186 (Part 1, Cohort S1) | A Single Dose MT-1186 (Part 1, Cohort S2) | A Single Dose MT-1186 (Part 1, Cohort S3) | A Single Dose MT-1186 (Part 1, Cohort S4) | A Single Dose MT-1186 (Part 1, Cohort S5) | A Single Dose MT-1186 (Part 1, Cohort S6) | A Single Dose MT-1186 (Part 1, Cohort S7) | Matching Placebo (a Single Dose Cohorts) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2) | Matching Placebo (Multiple Doses Cohorts) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 6 | 6 | 6 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 6 | 6 | 6 | 74
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 6 | 6 | 6 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0 | 0 | 8
  Asian (Japanese) | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 12 | 6 | 6 | 6 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (Aes) and Adverse Drug Reactions (ADRs)
Time Frame: Day 1 to 8 in Part 1, up to 12 days in Part 2
Population: The trial is divided into 2 phases (a single and multiple-dose). A single-dose study included 8 cohorts (total of 56 subjects), with 42 (6x7) subjects receiving MT-1186, and 14 (2x7) receiving the placebo. Multiple-dose study included 2 cohorts (total of 18 subjects), with 12 (6x2) receiving MT-1186, and 6 (3x2) receiving the placebo for 5 days. Since Cohort S3-1 and S3-2 are crossover cohort, the 5 subjects in Cohort S3-2 are overlapped (total of 79 subjects).
Measure: Count of Participants; unit: Participants
Groups:
- A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1): Healthy Japanese male subjects receive a single dose of MT-1186 60 mg solution under fasted condition.
- A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2): Healthy Japanese male subjects receive a single dose of MT-1186 120 mg suspension under fasted condition.
- A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1): Healthy Japanese male subjects receive a single dose of MT-1186 200 mg with fasted condition under period 1.
- A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2): Healthy Japanese male subjects receive a single dose of MT-1186 200 mg under fed condition in period 2 with washout period at least 4-day.
- A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4): Healthy Japanese male subjects receive a single dose of MT-1186 300 mg suspension with xanthan under fasted condition.
- A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5): Healthy Japanese male subjects receive a single dose of MT-1186 300 mg suspension under fasted condition.
- A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6): Healthy Japanese male subjects receive a single dose of MT-1186 30 mg solution under fasted condition.
- A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7): Healthy Caucasian male subjects receive a single dose of MT-1186 200 mg suspension under fasted condition.
- Matching Placebo Under Fasted Condition (a Sngle Dose Cohorts): Healthy Japanese/Caucasian male subjects receive a single dose of matching placebo.
- Multiple Doses MT-1186 (Part 2, Cohort M1): Healthy Japanese male subjects receive multiple doses of MT-1186 120 mg suspension under fasted condition.
- Multiple Doses MT-1186 (Part 2, Cohort M2): Healthy Japanese male subjects receive multiple doses of MT-1186 200 mg suspension under fasted condition.
- Matching Placebo (Multiple Doses Cohorts): Healthy Japanese male subjects receive multiple doses of matching placebo under fasted condition.
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Matching Placebo Under Fasted Condition (a Sngle Dose Cohorts) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2) | Matching Placebo (Multiple Doses Cohorts)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 14 | 6 | 6 | 6
Participants
  Participants with AEs | 0 | 2 | 3 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 1 | 1
  Participants with ADRs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC) of Unchanged Edaravone
Description: Area under the plasma concentration versus time curve from time zero up to 24 hours (AUC0-24) of unchanged edaravone.
Time Frame: Part 1: Pre-dose, 0.25, 0.5, 1.5, 2, 4, 6, 8, 12, 24, 36, 48 hrs post-dose, Part 2: Day 1 and 5 at pre-dose, 0.25, 0.5, 1.5, 2, 4, 6, 8, 12 hrs post-dose; Day 2 to 4 at pre-dose; Day 6 at 24 hrs post-dose on Day 5; Day 7 at 48 hrs post-dose on Day 5
Population: The trial is divided into 2 phases (a single and multiple-dose). A single-dose study included 8 cohorts (total of 56 subjects), with 42 (6x7) subjects receiving MT-1186, and 14 (2x7) receiving the placebo. Multiple-dose study included 2 cohorts (total of 18 subjects), with 12 (6x2) receiving MT-1186, and 6 (3x2) receiving the placebo for 5 days. Since Cohort S3-1 and S3-2 are crossover cohort, the 5 subjects in Cohort S3-2 are overlapped (59 patients receiving MT-1186).
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL
  AUC from time zero to 24 hour (AUC 0-24): Day 1 | 816 (231) | 2242 (911) | 6254 (1236) | 2443 (813) | 11319 (1053) | 9034 (2738) | 285 (113) | 4935 (1980) | 1917 (383) | 4133 (1260)
  AUC from time zero to 24 hour (AUC 0-24): Day 5, only Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  AUC from time zero to 24 hour (AUC 0-24): Day 5, only Part 2 |  |  |  |  |  |  |  |  | 2189 (516) | 4279 (1166)

3. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC) of Sulfate Conjugate
Description: Area under the plasma concentration versus time curve from time zero up to 24 hours (AUC0-24) of sulfate conjugate.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL
  AUC from time zero to 24 hour (AUC 0-24): Day 1 | 16251 (7143) | 30004 (6103) | 45666 (10447) | 38244 (4602) | 67693 (14170) | 68126 (15067) | 6709 (2171) | 44797 (16374) | 26132 (4083) | 39516 (3331)
  AUC from time zero to 24 hour (AUC 0-24): Day 5, only part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  AUC from time zero to 24 hour (AUC 0-24): Day 5, only part 2 |  |  |  |  |  |  |  |  | 24578 (4186) | 39102 (4208)

4. Primary Outcome: Area Under the Concentration Versus Time Curve (AUC) of Glucuronide Conjugate
Description: Area under the plasma concentration versus time curve from time zero up to 24 hours (AUC0-24) of glucuronide conjugate.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL
  AUC from time zero to 24 hour (AUC 0-24):Day 1 | 2360 (648) | 4815 (910) | 8146 (1275) | 7406 (1368) | 14403 (1557) | 12499 (3457) | 1201 (454) | 8038 (1898) | 4806 (509) | 7932 (1190)
  AUC from time zero to 24 hour (AUC 0-24): Day 5, only part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  AUC from time zero to 24 hour (AUC 0-24): Day 5, only part 2 |  |  |  |  |  |  |  |  | 4698 (499) | 8059 (1278)

5. Primary Outcome: Maximum Plasma Concentration (Cmax) of Unchanged Edaravone
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  Day 1 | 755 (356) | 1735 (738) | 4933 (1268) | 899 (464) | 8805 (933) | 5426 (2496) | 208 (112) | 3692 (1529) | 1953 (838) | 3855 (1676)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 2308 (941) | 4092 (1715)

6. Primary Outcome: Maximum Plasma Concentration (Cmax) of Sulfate Conjugate
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  Day 1 | 5481 (2337) | 9108 (2104) | 12190 (2087) | 7324 (743) | 14590 (2102) | 14080 (4787) | 2913 (870) | 11510 (2502) | 7318 (612) | 10830 (2346)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 7402 (954) | 11200 (1744)

7. Primary Outcome: Maximum Plasma Concentration (Cmax) of Glucuronide Conjugate
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL
  Day 1 | 1313 (378) | 2272 (279) | 3507 (158) | 1893 (358) | 5322 (958) | 3968 (912) | 750 (263) | 3361 (1183) | 2145 (356) | 3219 (666)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 2209 (156) | 3439 (428)

8. Primary Outcome: Part 2: Minimum Plasma Concentration at Steady State (Ctrough, ss)
Time Frame: Part 2: Day 1 and 5 at pre-dose, 0.25, 0.5, 1.5, 2, 4, 6, 8, 12 hrs post-dose; Day 2 to 4 at pre-dose; Day 6 at 24 hrs post-dose on Day 5; Day 7 at 48 hrs post-dose on Day 5
Population: The trial is divided into 2 phases (a single and multiple-dose). A single-dose study included 8 cohorts (S3-1 and S3-2 are crossover cohort, total of 56 subjects), with 42 (6x7) subjects receiving MT-1186, and 14 (2x7) receiving the placebo. Multiple-dose study included a total of 2 cohorts (total of 18 subjects), with 12 (6x2) receiving MT-1186, and 6 (3x2) receiving the placebo for 5 days.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6
ng/mL
  Unchanged Edaravone | 2.34 (0.30) | 3.79 (0.80)
  Sulfate conjugate | 32.91 (9.01) | 49.98 (11.22)
  Glucuronide conjugate | 2.69 (0.30) | 5.48 (1.90)

9. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Unchanged Edaravone
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
h
  Day 1 | 0.3 (0.1) | 0.4 (0.1) | 0.4 (0.1) | 1.4 (1.6) | 0.6 (0.3) | 0.8 (0.4) | 0.4 (0.1) | 0.6 (0.3) | 0.4 (0.1) | 0.4 (0.1)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 0.4 (0.1) | 0.4 (0.1)

10. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Sulfate Conjugate
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
h
  Day 1 | 0.6 (0.2) | 0.8 (0.3) | 1.0 (0.0) | 1.3 (0.5) | 1.3 (0.3) | 1.4 (0.4) | 0.5 (0.3) | 0.9 (0.4) | 0.8 (0.3) | 0.9 (0.2)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 0.8 (0.3) | 0.8 (0.3)

11. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Glucuronide Conjugate
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
h
  Day 1 | 0.5 (0.3) | 0.6 (0.2) | 0.6 (0.2) | 1.2 (0.6) | 1.0 (0.3) | 1.1 (0.4) | 0.5 (0.3) | 0.9 (0.4) | 0.7 (0.3) | 0.6 (0.2)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 0.6 (0.2) | 0.7 (0.3)

12. Primary Outcome: Terminal Elimination Half-life (t1/2) of Unchanged Edaravone
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
h
  Day 1 | 3.2 (0.9) | 5.1 (1.5) | 9.1 (2.4) | 5.2 (1.7) | 11.8 (4.) | 9.1 (3.3) | 2.4 (0.7) | 6.5 (1.7) | 4.6 (0.4) | 4.2 (0.2)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 8.7 (3.2) | 12.4 (1.9)

13. Primary Outcome: Terminal Elimination Half-life (t1/2) of Sulfate Conjugate
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
h
  Day 1 | 7.9 (2.6) | 7.3 (2.6) | 5.9 (1.7) | 5.1 (1.3) | 6.0 (1.6) | 4.9 (0.3) | 5.2 (0.6) | 6.4 (2.6) | 3.7 (0.2) | 3.4 (0.3)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 6.2 (0.4) | 6.8 (1.0)

14. Primary Outcome: Terminal Elimination Half-life (t1/2) of Glucuronide Conjugate
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
h
  Day 1 | 3.4 (1.1) | 3.2 (0.9) | 4.3 (0.7) | 3.8 (0.9) | 5.9 (1.4) | 4.8 (0.5) | 2.8 (0.9) | 4.7 (1.2) | 3.5 (0.2) | 3.2 (0.4)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 3.9 (0.3) | 5.2 (2.0)

15. Primary Outcome: Lambda-z of Unchanged Edaravone
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
1/h
  Day 1 | 0.23 (0.05) | 0.14 (0.03) | 0.08 (0.02) | 0.14 (0.04) | 0.07 (0.02) | 0.08 (0.02) | 0.31 (0.11) | 0.11 (0.03) | 0.15 (0.01) | 0.17 (0.01)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 0.09 (0.03) | 0.06 (0.01)

16. Primary Outcome: Lambda-z of Sulfate Conjugate
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
1/h
  Day 1 | 0.10 (0.03) | 0.11 (0.04) | 0.12 (0.02) | 0.14 (0.03) | 0.12 (0.03) | 0.14 (0.01) | 0.14 (0.02) | 0.12 (0.03) | 0.19 (0.01) | 0.20 (0.02)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 0.11 (0.01) | 0.10 (0.02)

17. Primary Outcome: Lambda-z of Glucuronide Conjugate
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
1/h
  Day 1 | 0.23 (0.09) | 0.23 (0.07) | 0.17 (0.03) | 0.19 (0.05) | 0.12 (0.02) | 0.15 (0.01) | 0.27 (0.07) | 0.16 (0.04) | 0.20 (0.01) | 0.22 (0.03)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 0.18 (0.01) | 0.15 (0.05)

18. Primary Outcome: Mean Residence Time (MRT) of Unchanged Edaravone
Time Frame: Part 1: Pre-dose, 0.25, 0.5, 1.5, 2, 4, 6, 8, 12, 24, 36, 48 hrs post-dose Part 2: Day 1 and 5 at pre-dose, 0.25, 0.5, 1.5, 2, 4, 6, 8, 12 hrs post-dose; Day 2 to 4 at pre-dose; Day 6 at 24 hrs post-dose on Day 5; Day 7 at 48 hrs post-dose on Day 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
h
  Day 1 | 1.92 (0.46) | 2.07 (0.26) | 1.98 (0.15) | 3.41 (0.62) | 2.14 (0.20) | 2.42 (0.45) | 2.02 (0.20) | 2.02 (0.32) | 1.94 (0.15) | 1.90 (0.26)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 2.17 (0.24) | 2.28 (0.37)

19. Primary Outcome: Apparent Total Clearance (CL/F) of Unchanged Edaravone
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- A Single Dose MT-1186 (Part 1, Cohort S6): Healthy Japanese male subjects receive a single dose of MT-1186 30 mg solution under fasted condition.
- Multiple Doses MT-1186 (Part 2, Cohort M1): Healthy Japanese male subjects receive multiple doses of MT-1186 200 mg suspension at 30 min before breakfast.
- Multiple Doses MT-1186 (Part 2, Cohort M2): Healthy Japanese male subjects receive multiple doses of matching placebo at 30 min before breakfast.
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
L/h
  Day 1 | 79.77 (26.21) | 60.29 (22.90) | 32.73 (6.42) | 87.07 (22.96) | 26.42 (2.30) | 36.11 (13.62) | 119.41 (43.64) | 46.72 (20.27) | 64.51 (11.64) | 53.40 (20.46)
  Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Day 5 |  |  |  |  |  |  |  |  | 57.64 (14.54) | 50.74 (18.08)

20. Primary Outcome: Apparent Distribution Volume at Elimination Phase (Vz/F) and Apparent Distribution Volume at Steady State (Vss/F) of Unchanged Edaravone
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S1) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S3-1) | A Single Dose MT-1186 Under Fed Condition(Part 1, Cohort S3-2) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S7) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2)
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 6 | 6
L
  Vz/F (Part 1), Vss/F (Part 2): Day1 | 348.98 (87.82) | 422.67 (126.97) | 426.49 (130.84) | 620.73 (139.24) | 457.99 (188.01) | 457.37 (175.69) | 384.51 (96.92) | 408.95 (121.29) | 126.41 (29.65) | 105.90 (57.04)
  Vss/F (only Part 2): Day 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
  Vss/F (only Part 2): Day 5 |  |  |  |  |  |  |  |  | 125.94 (40.36) | 121.32 (66.83)

21. Secondary Outcome: Change of Heart Rate (HR) From Baseline
Description: Holter ECG data were recorded in part 1, Cohorts S4, S5, and S6. Baseline is calculated as average HR from 0.75, 0.5, and 0.25 hours pre-dose.
Time Frame: 0.75, 0.5, and 0.25 hours pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose.
Population: Pharmacodynamic data were collected in Cohort S4, S5 and S6 with 18 (6x3 subjects receiving MT-1186), and 6 (2x3) receiving the placebo of Part 1.
Measure: Least Squares Mean (Standard Error); unit: bpm
Groups:
- Matching Placebo (a Sngle Dose Cohorts: Healthy Japanese male subjects receive a single dose of matching placebo.
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | Matching Placebo (a Sngle Dose Cohorts
Number analyzed (Participants) | 6 | 6 | 6 | 6
bpm
  0.25h | 1.8 (0.91) | -1.2 (0.91) | 1.8 (0.96) | -0.2 (0.92)
  0.5h | -0.2 (1.01) | 0.2 (1.01) | 1.3 (1.06) | 1.2 (1.02)
  1h | -0.1 (1.28) | -1.7 (1.28) | 0.2 (1.34) | -0.2 (1.29)
  1.5h | -1.2 (1.00) | -0.3 (1.00) | 0.2 (1.04) | -0.1 (1.01)
  2h | -0.1 (0.95) | 0.4 (0.95) | 0.9 (0.99) | -0.1 (0.96)
  4h | -0.7 (1.36) | -1.6 (1.36) | -0.1 (1.42) | -1.5 (1.37)
  6h | 3.2 (1.88) | 6.4 (1.87) | 3.8 (1.96) | 3.8 (1.89)
  8h | 4.4 (1.72) | 4.1 (1.72) | 6.2 (1.80) | 3.4 (1.74)
  12h | 1.9 (2.07) | 10.1 (2.07) | 7.6 (2.16) | 4.6 (2.09)
  24h | 1.3 (1.54) | 1.7 (1.54) | 2.2 (1.61) | -1 (1.55)
  36h | 8.1 (3.07) | 9.9 (3.06) | 13.2 (3.21) | 5.7 (3.10)
  48h | 4.3 (2.51) | 8.2 (2.51) | 8.4 (2.62) | 2.4 (2.53)

22. Secondary Outcome: Change of PR Interval (PR) From Baseline
Description: as for outcome 21
Time Frame: 0.75, 0.5, and 0.25 hours pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose.
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | Matching Placebo (a Sngle Dose Cohorts
Number analyzed (Participants) | 6 | 6 | 6 | 6
msec
  0.25h | -6.8 (1.91) | -3.3 (1.99) | -5.7 (1.92) | -4.5 (2.06)
  0.5h | -4.2 (1.35) | 0.1 (1.40) | -2.4 (1.36) | -3.4 (1.45)
  1h | -4.2 (1.68) | 2.1 (1.74) | -4.0 (1.68) | -4.7 (1.80)
  1.5h | -5.2 (2.23) | 0.0 (2.31) | -4.8 (2.24) | -5.3 (2.40)
  2h | -5.9 (1.90) | -0.8 (1.97) | -4.5 (1.91) | -5.9 (2.05)
  4h | -3.0 (2.64) | -3.0 (2.74) | -5.3 (2.66) | -5.4 (2.85)
  6h | -5.5 (1.91) | -9.6 (1.98) | -6.3 (1.92) | -6.6 (2.06)
  8h | -11.6 (2.60) | -9.0 (2.70) | -9.9 (2.62) | -11.9 (2.80)
  12h | -6.6 (3.91) | -12.0 (4.06) | -9.0 (3.93) | -11.8 (4.21)
  24h | -2.1 (2.62) | -1.6 (2.72) | -8.9 (2.63) | -1.1 (2.82)
  36h | -5.7 (3.77) | -6.8 (3.91) | -6.2 (3.78) | -9.5 (4.06)
  48h | -3.3 (2.63) | 0.6 (2.73) | -3.2 (2.64) | -5.4 (2.83)

23. Secondary Outcome: Change of QTcF Interval (QTcF) From Baseline
Description: as for outcome 21
Time Frame: 0.75, 0.5, and 0.25 hours pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose.
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | Matching Placebo (a Sngle Dose Cohorts
Number analyzed (Participants) | 6 | 6 | 6 | 6
msec
  0.25h | 2.0 (1.60) | 0.7 (1.60) | 1.6 (1.63) | 0.8 (1.71)
  0.5h | -2.2 (1.32) | 1.1 (1.31) | -3.8 (1.34) | -4.9 (1.41)
  1h | 0.3 (2.02) | -0.1 (2.02) | -4.7 (2.06) | 0.5 (2.17)
  1.5h | -5.2 (2.23) | 2.7 (1.68) | -1.9 (1.71) | -5.3 (2.40)
  2h | 1.2 (1.68) | 1.5 (2.34) | -5.1 (2.39) | 0.8 (1.80)
  4h | 2.3 (2.85) | -0.9 (2.85) | 1.4 (2.90) | 0.7 (3.06)
  6h | -5.7 (2.96) | -2.9 (2.96) | -7.6 (3.01) | -2.4 (3.18)
  8h | -5.3 (2.62) | -2.9 (2.62) | -7.0 (2.66) | -6.9 (2.81)
  12h | -2.3 (2.42) | -4.0 (2.42) | -3.1 (2.47) | -3.3 (2.6)
  24h | 2.0 (2.42) | -1.2 (2.42) | -5.7 (2.46) | -3.1 (2.60)
  36h | -3.0 (2.96) | -5.0 (2.96) | -5.1 (3.01) | -1.4 (3.18)
  48h | -1.0 (3.22) | -1.5 (3.22) | -4.4 (3.28) | -0.1 (3.46)

24. Secondary Outcome: Change of QRS Duration (QRS) From Baseline
Description: Holter ECG data were recorded in part 1, Cohorts S4, S5, and S6.
Time Frame: 0.75, 0.5, and 0.25 hours pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 24, 36, and 48 hours post-dose.
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: msec
Arm/Group | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S4) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S5) | A Single Dose MT-1186 Under Fasted Condition (Part 1, Cohort S6) | Matching Placebo (a Sngle Dose Cohorts
Number analyzed (Participants) | 6 | 6 | 6 | 6
msec
  0.25h | -0.7 (0.85) | -0.4 (0.84) | 0.4 (0.87) | -2.0 (0.88)
  0.5h | -0.3 (0.77) | -0.8 (0.77) | -0.5 (0.80) | -1.6 (0.80)
  1h | -0.3 (0.70) | -1.5 (0.69) | 0.5 (0.72) | -1.4 (0.72)
  1.5h | -0.4 (0.70) | -0.7 (0.80) | 0.4 (0.83) | -1.4 (0.72)
  2h | -1.5 (0.98) | -0.5 (0.98) | 0.2 (1.01) | -2.7 (1.02)
  4h | -0.5 (1.36) | -2.1 (1.36) | -0.4 (1.41) | -0.5 (1.42)
  6h | -0.3 (1.31) | 1.1 (1.31) | -0.8 (1.36) | 0.7 (1.37)
  8h | -1.2 (1.50) | 0.0 (1.50) | -2.4 (1.55) | -1.3 (1.57)
  12h | 0.4 (1.71) | -2.1 (1.71) | -2.0 (1.77) | 0.0 (1.78)
  24h | -0.9 (1.26) | -2.2 (1.25) | -1.4 (1.30) | -1.2 (1.31)
  36h | -0.2 (1.76) | -1.5 (1.75) | -2.4 (1.81) | 0.4 (1.83)
  48h | -1.7 (1.18) | -1.5 (1.17) | -1.4 (1.22) | -0.1 (1.23)

ADVERSE EVENTS:
Time Frame: 8 days in part 1, 12 days in part 2
Arm/Group | A Single Dose MT-1186 (Part 1, Cohort S1) | A Single Dose MT-1186 (Part 1, Cohort S2) | A Single Dose MT-1186 (Part 1, Cohort S3) | A Single Dose MT-1186 (Part 1, Cohort S4) | A Single Dose MT-1186 (Part 1, Cohort S5) | A Single Dose MT-1186 (Part 1, Cohort S6) | A Single Dose MT-1186 (Part 1, Cohort S7) | Matching Placebo (a Single Dose Cohorts) | Multiple Doses MT-1186 (Part 2, Cohort M1) | Multiple Doses MT-1186 (Part 2, Cohort M2) | Matching Placebo (Multiple Doses Cohorts)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 3/6 | 0/6 | 1/6 | 1/6 | 2/6 | 2/14 | 2/6 | 1/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A Single Dose MT-1186 (Part 1, Cohort S1) (N=6) | A Single Dose MT-1186 (Part 1, Cohort S2) (N=6) | A Single Dose MT-1186 (Part 1, Cohort S3) (N=6) | A Single Dose MT-1186 (Part 1, Cohort S4) (N=6) | A Single Dose MT-1186 (Part 1, Cohort S5) (N=6) | A Single Dose MT-1186 (Part 1, Cohort S6) (N=6) | A Single Dose MT-1186 (Part 1, Cohort S7) (N=6) | Matching Placebo (a Single Dose Cohorts) (N=14) | Multiple Doses MT-1186 (Part 2, Cohort M1) (N=6) | Multiple Doses MT-1186 (Part 2, Cohort M2) (N=6) | Matching Placebo (Multiple Doses Cohorts) (N=6)
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT04481750/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT04481750/SAP_001.pdf